CLINICAL TRIAL: NCT00728455
Title: Single Subcutaneous Dose Rising Study to Investigate the Safety, Tolerability, Efficacy and Pharmacokinetics of NNC 0070-0002-0349 in Overweight/Obese Male Subjects
Brief Title: Examination of the Safety and Tolerability of NNC 0070-0002-0349 in Overweight/Obese Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9112-1905
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- A (Experimental)
  Interventions: Drug: NNC 0070-0002-0349; Drug: placebo
- B (Experimental)
  Interventions: Drug: NNC 0070-0002-0349; Drug: placebo
- C (Experimental)
  Interventions: Drug: NNC 0070-0002-0349; Drug: placebo
- D (Experimental)
  Interventions: Drug: NNC 0070-0002-0349; Drug: placebo
- E (Experimental)
  Interventions: Drug: NNC 0070-0002-0349; Drug: placebo

INTERVENTIONS:
Drug: NNC 0070-0002-0349 — Dose level 1: (6 subjects active, 2 subjects placebo). Subjects administered NNC 0070-0002-0349 will receive a subcutaneous injection. Subjects in the first 3 dose groups will receive two injections: one of randomized treatment (drug or placebo) and placebo
  Arms: A
Drug: NNC 0070-0002-0349 — Dose level 2: (6 subjects active, 2 subjects placebo). Subjects administered NNC 0070-0002-0349 will receive a subcutaneous injection. Subjects in the first 3 dose groups will receive two injections: one of randomized treatment (drug or placebo) and placebo
  Arms: B
Drug: NNC 0070-0002-0349 — Dose level 3: (6 subjects active, 2 subjects placebo). Subjects administered NNC 0070-0002-0349 will receive a subcutaneous injection. Subjects in the first 3 dose groups will receive two injections: one of randomized treatment (drug or placebo) and placebo
  Arms: C
Drug: NNC 0070-0002-0349 — Dose level 4 for s.c. injection (6 subjects active, 2 subjects placebo)
  Arms: D
Drug: NNC 0070-0002-0349 — Dose level 5 for s.c. injection (6 subjects active, 2 subjects placebo)
  Arms: E
Drug: placebo — Dose level 1: NNC 0070-0002-0349 placebo. Subjects administered placebo will receive a subcutaneous injection. Subjects in the first 3 dose groups will receive two injections: one of randomized treatment (drug or placebo) and placebo
  Arms: A
Drug: placebo — Dose level 2: NNC 0070-0002-0349 placebo. Subjects administered placebo will receive a subcutaneous injection. Subjects in the first 3 dose groups will receive two injections: one of randomized treatment (drug or placebo) and placebo
  Arms: B
Drug: placebo — Dose level 3: NNC 0070-0002-0349 placebo. Subjects administered placebo will receive a subcutaneous injection. Subjects in the first 3 dose groups will receive two injections: one of randomized treatment (drug or placebo) and placebo
  Arms: C
Drug: placebo — Dose level 4: NNC 0070-0002-0349 placebo for s.c. injection
  Arms: D
Drug: placebo — Dose level 5: NNC 0070-0002-0349 placebo for s.c. injection
  Arms: E

SUMMARY:
This trial will be conducted in the United States of America (USA). The aim of this clinical trial is to investigate whether NNC 0070-0002-0349 is safe and well tolerated.

Groups of eight subjects will be administered subcutaneous injections of NNC 0070-0002-0349 or placebo on Day 1 beginning with a low dose; after which laboratory and vital sign data as well as subject reported adverse events will be evaluated. If safe to proceed, the next group of subjects will be given a higher dose and the safety evaluation performed again before proceeding. In total, 5 dose levels will be evaluated.

Subjects will be administered a dose and remain in the clinic until the morning of Day 8 after dosing and vital signs and safety labs as well as blood drawn for pharmacokinetic samples taken. Subjects will return to the clinic on Days 10, 12, 14, 16, 18 and 22 for repeat blood draws and safety labs. Day 22 is the final study visit.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than 27.0 and less than 35.0 kg/m2

Exclusion Criteria:

* Systolic blood pressure greater than 140 mm Hg or diastolic greater than 90 mm Hg
* Depression or suicidal thoughts (Scoring on Patient Health Questionnaire-9-item)
* Eating disorders
* Unusual diets or eating habits
* Dieting, use of diet drugs or obesity surgery
* Diabetes history or abnormal fasting glucose

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability (adverse events, vital signs, blood chemistry, physical examination, ECG) | Including screening and evaluation: after approx. 7 weeks

SECONDARY OUTCOMES:
AUC (area under the curve) | 21 days following dosing
Maximum plasma concentration | 21 days following dosing
Time to maximum plasma concentration | 21 days following dosing
Half life | 21 days following dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com